CLINICAL TRIAL: NCT05463224
Title: Lazertinib for NSCLC Harboring Activating EGFR Mutations in TKI naïve Patients: A Single-arm, Phase II Single-center Trial
Brief Title: Lazertinib for NSCLC Harboring Activating EGFR Mutations in TKI naïve Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Se-Hoon Lee (Other)
Responsible Party: Sponsor-Investigator, Se-Hoon Lee, M.D, Ph.D. Principal Investigator, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-09-029
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: NSCLC
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Intervention Model Description: A single-arm, phase II single-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lazertinib group (Experimental): Lazertinib 240mg daily (1 cycle of 21 days)
  Interventions: Drug: Lazertinib group

INTERVENTIONS:
Drug: Lazertinib group — Lazertinib 240mg, Once, po, daily (1 cycle of 21 days)
  Other Names: Leclaza

SUMMARY:
The primary objective is to evaluate the efficacy/safety of lazertinib and to explore the resistance mechanism of lazertinib as first-line in patients with NSCLC harboring activating EGFR mutations.

DETAILED DESCRIPTION:
As the 3rd generation EGFR TKI become a standard treatment option for the 1st line therapy in EGFR mutated patients, necessity for evaluating resistant mechanism to determine the matched subsequent therapeutic option has been highlighted. The idea of understanding the exact resistance mechanism to 1st line 3rd generation EGFR TKI treatment is emphasized based on the observation that resistance mechanism is different based on osimertinib used as 1st line or 2nd line treatment.6,7 Although resistance mechanisms to lazertinib in patients with prior EGFR TKI treatment have been studied, there are no current data available regarding the resistance mechanism after first-line lazertinib treatment.

Based on this observation, PI designed this study to elucidate the efficacy/safety of Lazertinib and to explore resistance mechanisms of 1st line lazertinib treatment in NSCLC patients with activating EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer which is not amenable to treatment with a curative aim (e.g. surgery or radiation). Patients who underwent curative intent surgery or definitive CRT and experience recurrence after 6 months are eligible.
* Stage IIIC or IV by AJCC 8th edition
* Confirmed EGFR mutations (exon 19 deletion, L858R)(The result from both cell-free DNA or tissue-based DNA from the local test is allowed.)
* Age of 19 or more.
* Performance status of Eastern Cooperative Oncology Group 0 to 2.
* Expected minimum life expectancy of 12 weeks
* Adequate organ function.

  * Available to provide the adequate tissue and blood for the genomic tests- At least 15 unstained slide and 20 cc of blood at baseline (mandatory) and disease progression.
* Agreed to perform re-biopsy at the timepoint of disease progression.
* At least two weeks after the chemotherapy
* Female subjects must either be of non-reproductive potential
* Subject willing and able to comply with the protocol
* Signed written informed consent

Exclusion Criteria:

* Previously treatment with any kind of EGFR TKI (Previously chemotherapy treated patients is allowed)
* Any concurrent and/or other active malignancy that has required systemic treatment within 2 years of first dose of study drug. (allowed for participation if investigator decided that previous malignancy is cured and not need for any additional treatment)
* Uncontrolled central nervous system metastases- patient with asymptomatic brain metastases or CNS symptom manageable with TKI and evaluated by investigator can be enrolled.
* Spinal cord compression, leptomeningeal carcinomatosis
* Uncontrolled systemic illness, including uncontrolled hypertension, active bleeding, or active infection
* Radiotherapy with a wide field of radiation within 2 weeks or radiotherapy with a limited field of radiation (localized radiotherapy or gamma knife surgery) for palliation within 1 week
* Any unresolved toxicities from prior therapy, greater than CTCAE grade 1
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms
* No measurable lesion
* Unable to swallow the product due to refractory nausea, vomiting or chornic gastrointestinal disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | through study completion, an average of 18.0 month
  C1D1 until the date of objective disease progression or death
Resistance mechanism analysis | Screening, Discontiunuation Visit
  The mutation profile of baseline and at the timepoint of resistance will be evaluated using tissue and cfDNA

SECONDARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 18.0 month
  as the percentage of patients with measurable disease with at least one visit response of complete response (CR) or partial response (PR)
Duration of Response (DoR) | through study completion, an average of 18.0 month
  as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first
Disease control rate (DCR) | through study completion, an average of 18.0 month
  as the percentage of patients who have a best overall response of CR or PR or stable disease (SD at ≥ 6 weeks, prior to any PD event)
Overall survival (OS) | through study completion, an average of 18.0 month
  s the time from the date of C1D1 until the date of death due to any cause
intracranial PFS (iPFS) | through study completion, an average of 18.0 month
  as the time from C1D1 until the date of objective intracranial disease progression or death whichever comes first in patients for the iFAS
intracranial ORR (iORR) | through study completion, an average of 18.0 month
  as the percentage of patients who have at least 1 CR or PR in intracranial lesion, according to RECIST v1.1 prior to disease progression in patients who have at least one measurable intracranial lesion at baseline
intracranial DCR (iDCR) | through study completion, an average of 18.0 month
  as the percentage of patients who have a best intracranial overall response of CR or PR or SD in patients who have at least one measurable intracranial lesion at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnamgu, South Korea

IPD SHARING:
Plan to Share IPD: No